CLINICAL TRIAL: NCT04721782
Title: Assessment of Effects of Maternal Smoking on Fetal Liver Circulation With Ultrasonography
Brief Title: Effects of Maternal Smoking on Fetal Liver Circulation
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Bezmialem Vakif University (Other)
Collaborators: Maternal Fetal Medicine and Perinatology Society of Turkey (Unknown)
Responsible Party: Principal Investigator, Mehmet Serdar Kutuk, Associate Professor, Bezmialem Vakif University
Other Study IDs: 06/109
Record Dates: First submitted 2020-12-03; First posted 2021-01-25 (Actual); Last update posted 2021-01-25 (Actual); Status verified 2021-01

CONDITIONS: Smoking, Cigarette; Maternal Exposure; Ultrasound; Fetal; Circulation; Liver
Keywords: Cotinine; Carbon monoxide; Smoking; Fetal; Liver circulation
MeSH Terms: conditions — Cigarette Smoking; Persistent Fetal Circulation Syndrome; Smoking | interventions — Smoking Devices

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 20 Weeks

GROUPS / COHORTS (2):
- otherwise healthy, smoking, singleton pregnant women between 24- 36 weeks: Fetal liver circulation will be evaluated with doppler ultrasound, The degree of maternal smoking will be assessed by measuring urine cotinine and exhaled carbon monokside levels
  Interventions: Other: smoking
- otherwise healthy, non-smoking, singleton pregnant women between 24- 36 weeks: Fetal liver circulation will be evaluated with doppler ultrasound, The degree of maternal smoking will be assessed by measuring urine cotinine and exhaled carbon monokside levels

INTERVENTIONS:
Other: smoking — to assess the effect of smoking of fetal liver circulation with prenatal Doppler Ultrasonography
  Groups: otherwise healthy, smoking, singleton pregnant women between 24- 36 weeks

SUMMARY:
According to the hypothesis of this study presented, the effects of smoking on the fetus can be determined by the liver circulation and hepatic metabolism. The basic assumption of this project is; Compensatory and pathological findings can be seen in the fetal liver circulation in babies of mothers who smoke and the findings can be valuable in predicting the direction of fetal development (growth retardation or normal development). In this study, the flow and shunt amounts in the fetal hepatic vessels in normal and smoking pregnant women will be calculated with the help of Doppler US.

DETAILED DESCRIPTION:
Smoking is an agent that negatively affects of uteroplacental circulation and fetal development due to the chemical substances it contains, especially carbon monoxide and nicotine. According to the hypothesis of this study presented, the effects of smoking on the fetus can be determined by the liver circulation and hepatic metabolism. The basic assumption of this project is; Compensatory and pathological findings can be seen in the fetal liver circulation in babies of mothers who smoke and the findings can be valuable in predicting the direction of fetal development (growth retardation or normal development). In this study, the flow and shunt amounts in the fetal hepatic vessels in normal and smoking pregnant women will be calculated with the help of Doppler US.Therefore, we try to delineate pathological circulatory pattern in these fetuses and shed light to the mechanism of smoking-induced abnormal fetal development. In addition, the effects of other maternal demographic factors, cigarette amount, cotinine and expiratory carbon monoxide levels (or any correlation between them) on hepatic circulation and fetal development will be examined.

ELIGIBILITY:
Inclusion Criteria:

* singleton pregnancy
* smoking more than one cigarette in a day

Exclusion Criteria:

* fetal anomaly
* pregnant women with systemic disease
* younger than 18 years

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — pregnancy
Study Population: women who smoke during singleton pregnancy, without fetal anomaly and systemic disease
Sampling Method: Non-Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2020-07-07 (Actual); Primary Completion 2020-09-10 (Actual); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
Comparison of hepatic venous flow between smoking and non- smoking pregnant women | 24-36 weeks of pregnancy
  The evaluation of fetal flow parameters will be done with Voluson E6 and Philips EPIQ Elite ultrasound devices.
  In evaluations, diameters and the time avaraged flow velocities in intraabdominal umbilical vein, left portal vein, main portal vein and ductus venosus (DV) will be measured. The flow volumes will be calculated according to the specified formula and the venous flow of the right and left lobes of the liver and total venous flow of the liver will be determined, adjusted for estimated fetal weight and compared between groups.
  Flow Formulas; (QUV, QDV, QLPV, QPV):
  Total venous Hepatic Flow (Qhep)= (QUV-QDV) + QPV Flow to the left liver lobe(QLL)= QUV - (QDV + QleftPV) Flow to the right hepatic lobe (QrightLobe) = QPV + QleftPV

SECONDARY OUTCOMES:
The effect of maternal smoking on fetal growth | 24-36 weeks of pregnancy
  In the evaluation of fetal growth, fetal biometry (bipariatal diameter, head circumference, abdominal circumference, femur length) will be measured with ultrasound and estimated weight will be calculated with the headlock formula. The calculated weight will be compared with the appropriate (reference) normograms. Cases with estimated fetal weight (EFW) below 10 percentile will be considered as intrauterine growth retardation (IUGR).
  In both groups (smoking and non-smoking pregnant women) fetal biometry parameters will be measured and estimated fetal weight will be calculated.To be determined if maternal smoking has an effect on fetal growth retardation.
Sensitivity and specificity of maternal expiratory CO levels for detecting maternal smoking during pregnancy | 24-36 weeks of pregnancy
Normal references values of fetal umbilical venous and portal venous flow in Turkish Population | 24-36 weeks of pregnancy
  Doppler examination of the umbilical vein and portal vein in non-smokig pregnant women will determine the flow rate, flow volume and flow indexes in these vessels. In this way, it is planned to create a reference scale specific to the week of gestation for these parameters in healthy pregnant women in the Turkish population.

CONTACTS AND LOCATIONS:
Locations (1):
- Bezmialem Vakıf University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cnattingius S. The epidemiology of smoking during pregnancy: smoking prevalence, maternal characteristics, and pregnancy outcomes. Nicotine Tob Res. 2004 Apr;6 Suppl 2:S125-40. doi: 10.1080/14622200410001669187. PMID 15203816
- [Background] Kallen K. Maternal smoking during pregnancy and infant head circumference at birth. Early Hum Dev. 2000 Jun;58(3):197-204. doi: 10.1016/s0378-3782(00)00077-3. PMID 10936439
- [Background] Kiserud T. Fetal venous circulation--an update on hemodynamics. J Perinat Med. 2000;28(2):90-6. doi: 10.1515/JPM.2000.011. PMID 10875092